CLINICAL TRIAL: NCT02946502
Title: Prognostic Value of Dominant Hand Held Dynamometry in Mechanical Ventilation Weaning: a Prospective, Multicenter Study
Brief Title: Handgrip Strength Value in Predicting Mechanical Ventilation Weaning
Acronym: GRIPWEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P150948
Record Dates: First submitted 2016-10-18; First posted 2016-10-27 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Ventilator Weaning; Hand Strength; Respiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Handheld dynamometry (handgrip strength) (Experimental): All included patients will have a blinded evaluation of handgrip strength before weaning process.
  Interventions: Procedure: Handheld dynamometry (handgrip strength)

INTERVENTIONS:
Procedure: Handheld dynamometry (handgrip strength) — Patients will perform handgrip strength dynamometry through holding the device in their dominant hand with the maximum strength, with standardized arm and body positions, as well as incentives

SUMMARY:
The purpose of this study is to test the association between ICU acquired weakness as evaluated by dominant handheld dynamometry (handgrip) and the mechanical ventilation weaning outcome

DETAILED DESCRIPTION:
Previous studies have evidenced that Intensive Care Unit acquired peripheral muscle weakness may lead to delayed mechanical ventilation weaning (i.e difficult or prolonged weaning according to guidelines). Nevertheless, no study has ever tested the association between handgrip strength and extubation outcome. The investigators have generated the hypothesis that ICU acquired weakness, as tested by handgrip strength might be associated with extubation outcome. The investigators have planned to include 240 patients. Handgrip strength will be monitored, along with a full muscular assessment through Medical Research Council score by the attending physiotherapist. Physicians in charge of the patients will be blinded to these values and the weaning protocol will continue according to guidelines.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* under mechanical ventilation for at least 48 hours
* meeting readiness to wean criteria according to international guidelines
* with social security
* informed consent given by the patient or a proxy

Exclusion Criteria:

* baseline pre existing rheumatologic or neurologic condition preventing the patient to use the tested device
* confusion (as assessed by Confusion Assessment Method for the Intensive Care Unit )
* Patients whose extubation is a terminal extubation, or with prior decision not to resort a reintubation in case of post-extubation respiratory distress.
* known pregnancy
* Inability to deliver clear patient information (language barrier without an interpreter, for example)
* Participation in another intervention research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2017-01-17; Primary Completion 2019-11 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
extubation outcome according to handgrip strength value | 7 days
  Each mechanical ventilation weaning trial

SECONDARY OUTCOMES:
Association between handgrip strength and difficulty of weaning according to guidelines | 7 days
  Each mechanical ventilation weaning trial
Association between handgrip strength and cough strength as assessed through peak expiratory flow evaluated with a portable spirometer | 7 days
  Each mechanical ventilation weaning trial
Association between handgrip strength and maximal inspiratory strength during a brief inspiratory valve occlusion on the ventilator | 7 days
  Each mechanical ventilation weaning trial
Association between handgrip strength and peripheral muscular strength evaluated by the Medical Research Council score | 7 days
  Each mechanical ventilation weaning trial
Association between handgrip strength and the peripheral muscular strength evaluated by the Medical Research Council score. (Global score and its components) | 7 days
  Each mechanical ventilation weaning trial
Association between handgrip strength defined Intensive Care Unit acquired weakness and Intensive Care Unit and hospital length of stay | 18 months
Association between handgrip strength defined Intensive Care Unit acquired weakness and Intensive Care Unit and hospital survival | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Benjamin Sztrymf, Clamart, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cottereau G, Messika J, Megarbane B, Guerin L, da Silva D, Bornstain C, Santos M, Ricard JD, Sztrymf B. Handgrip strength to predict extubation outcome: a prospective multicenter trial. Ann Intensive Care. 2021 Oct 2;11(1):144. doi: 10.1186/s13613-021-00932-3. PMID 34601639